CLINICAL TRIAL: NCT06108726
Title: A Single-arm, Exploratory Clinical Trial Investigating the Efficacy of Local Envafolimab Injection Under Fiberoptic Bronchoscopy Combined With Chemotherapy in Non-small Cell Lung Cancer
Brief Title: A Study of Local Envafolimab Injection Combined With Chemotherapy in Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, xu xingxiang, Director, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xxingxiang
Record Dates: First submitted 2023-10-24; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: NSCLC
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- envafolimab plus chemotherapy (Experimental): Local injection of Envafolimab 5mg/kg plus platinum-based chemotherapy under fiberoptic bronchoscopy, Q2W.
  Interventions: Drug: Envafolimab Injection

INTERVENTIONS:
Drug: Envafolimab Injection — Local injection of Envafolimab 5mg/kg plus platinum-based chemotherapy under fiberoptic bronchoscopy, Q2W.
  Other Names: KN035

SUMMARY:
The aim of this single-arm, exploratory clinical study is to evaluate the safety and efficacy of local injection of envafolimab combined with chemotherapy in the first-line treatment of non-small cell lung cancer (NSCLC) patients, and to observe the changes of immune cells in the local immune microenvironment before and after immunotherapy, in order to find new indicators for immunotherapy evaluation.

DETAILED DESCRIPTION:
In this study, 16 patients with NSCLC were enrolled to explore the clinical effect of chemotherapy combined with local injection of Envafolimab. To determine whether the treatment of metastatic/recurrent NSCLC with Envafolimab is effective, and whether the treatment of Envafolimab combined with chemotherapy can prolong the PFS\OS of patients with NSCLC, and to screen for a more effective treatment mode for Chinese NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects volunteered to participate in the study, signed the informed consent form, and had good compliance;
* 2. ECOG≤2 ;
* 3.Life expectancy of ≥12 weeks；
* 4.Age ≥18 years;
* 5. Diagnosed by histological examination and/or cytology examination, and imaging evaluation (refer to RECIST 1.1) for advanced central NSCLC;
* 6. He had not received systemic chemotherapy previously.
* 7.Had at least one measurable tumor lesion according to RECIST v1.1；That is, in CT or MRI detection, the longest diameter of a single lesion is ≥10mm, or the lymph node is pathologically enlarged, and the short diameter of a single lymph node on CT scan is ≥15mm；
* 8.Have adequate organ function。

Exclusion Criteria:

* 1.This study was conducted five years prior to the initiation of treatment or concurrently with other malignant tumors.
* 2. Have family history of cancer.
* 3.had previously undergone any form treatment, such as surgery, chemotherapy, radiation therapy, etc.
* 4.Only individuals experiencing grade 1 or higher unmitigated toxic effects (excluding alopecia and fatigue) resulting from previous therapies were eligible for enrollment; neurologic toxicity needed to return to grade 1 or lower or baseline before participation.
* 5.Subjects with severe and/or uncontrollable disease progression；
* 6.Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
* 7.Pregnant or lactating women;
* 8.Other conditions considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | Up to 2 years
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate(ORR) | Up to 2 years
  ORR is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1
Progression free survival(PFS) | Up to 2 years
  Progression free survival (PFS) is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST v1.1.
Duration of response (DOR) | Up to 2 years
  DOR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Treatment related adverse events (TRAEs) | from first dose to 30 days post the last dose
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: xu X xiang, Doctor, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu People's Hospital, Suzhou, Jiangsu, China